CLINICAL TRIAL: NCT06939829
Title: A Prospective, Open-Label, Randomized Controlled, Multicenter Clinical Study on Continuous vs. Intermittent Infusion of Ceftazidime-Avibactam in Critically Ill Patients With Severe Infections
Brief Title: A Multicenter Clinical Study on the Continuous vs. Intermittent Infusion of Ceftazidime-Avibactam in Critically Ill Patients With Severe Infections
Acronym: AVIATOR
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jianfeng Xie, director, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025ZDSYLL022
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Patients With Critically Ill Infections
Keywords: Ceftazidime-Avibactam; Continuous versus Intermittent Infusion; clinical study
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the intermittent infusion group (Active Comparator): Ceftazidime-avibactam will be administered as 2.5 g q8h by intermittent infusion for 2 h, and the dosage could be adjusted according to the instructions.
  Interventions: Drug: treatment with CAZ-AVI
- the continuous infusion group (Experimental): After a loading dose of ceftazidime-avibactam, continuous infusion is administered, with the dose adjustment rules consistent with those of the intermittent infusion group.
  Interventions: Drug: treatment with CAZ-AVI

INTERVENTIONS:
Drug: treatment with CAZ-AVI — Randomize subjects to receive CAZ-AVI via either continuous infusion or intermittent infusion. The total daily dose and dosing interval should be determined according to the subject's body weight, renal function, and estimated drug clearance based on standard prescribing guidelines. Regardless of administration method, the same criteria for dose adjustment (including indications for modification and monitoring parameters) must be consistently applied to both control and experimental groups.

SUMMARY:
The objective of this study is to determine whether continuous infusion of ceftazidime-avibactam (CAZ-AVI) could improve clinical outcomes in critically ill patients compared with intermittent infusion.

DETAILED DESCRIPTION:
This study employs a prospective, open-label, randomized controlled, multicenter clinical trial design comparing "CAZ-AVI continuous infusion" versus "CAZ-AVI intermittent infusion," .The secondary objectives is to observe the clinical cure, Bacterial clearance, the probability of target attainment (PTA) of TDM. etc

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years old, male or female.
* Patients who are admitted to ICU wards.
* Patients clinically diagnosed with carbapenem-resistant organism (CRO) infections, and has been commenced on targeted therapy with ceftazidime-avibactam.
* One or more organ dysfunction criteria in the previous 24 hours i. MAP < 60 mmHg for at least 1 hour; ii. Vasopressors required for > 4 hours; iii. Respiratory support using supplemental high flow nasal prongs, continuous positive airway pressure, bilevel positive airway pressure or invasive mechanical ventilation for at least 1 hour.

iv. Serum creatinine concentration > 220 μmol/L or >2.49 mg/dL

Exclusion Criteria:

* Patient has a known allergy to ceftazidime-avibactam.
* Patient has received ceftazidime-avibactam for more than 48 hours during current infectious episode.
* Patient is in severe condition or expected to survive for no more than 48 hours.
* Patient who receives lung or heart transplant or stem cell transplant.
* Patient is known or suspected to be pregnant.
* Patient has previously been enrolled in the current study.
* Other conditions which are regarded as inappropriate for enrollment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
90-day all cause mortality | from randomization to day 90
  the proportion of subjects who die within 90 days after randomization to the number of subjects in each group

CONTACTS AND LOCATIONS:
Overall Officials: Feng jian Xie, MD, Study Chair — Department of Critical Care Medicine, Zhongda Hospital, School of Medicine, Southeast University

IPD SHARING:
Plan to Share IPD: No